CLINICAL TRIAL: NCT04778787
Title: Impact of Sodium-glucose Cotransporter Type 2 Inhibitors on the Course of Cardiorenal Syndrome in Acute Decompensation of Chronic Heart Failure
Brief Title: Sodium-glucose Cotransporter Type 2 Inhibitors for Acute Cardiorenal Syndrome Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10773100889666
Record Dates: First submitted 2021-02-17; First posted 2021-03-03 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-03

CONDITIONS: Congestive Heart Failure
Keywords: heart failure; decompensation; gliflozins; kidneys
MeSH Terms: conditions — Heart Failure | interventions — Sodium Potassium Chloride Symporter Inhibitors; Vasodilator Agents; Digoxin; Vasoconstrictor Agents; dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): The intervention group includes patients with decompensated chronic heart failure. The diagnosis will be made according to the criteria described above
  Interventions: Drug: Standard list of drugs used for acute decompensation of CHF (loop diuretics, vasodilators, digoxin, inotropic agents, vasopressors), plus dapagliflozin (Forxiga; MP-002596)
- the control group (Experimental): The control group will be identical to the main group.
  Interventions: Drug: Standard list of drugs used for acute decompensation of CHF (loop diuretics, vasodilators, digoxin, inotropic agents, vasopressors), plus dapagliflozin (Forxiga; MP-002596)

INTERVENTIONS:
Drug: Standard list of drugs used for acute decompensation of CHF (loop diuretics, vasodilators, digoxin, inotropic agents, vasopressors), plus dapagliflozin (Forxiga; MP-002596) — Patients will receive dapagliflozin at a dose of 10 mg daily during hospitalization in addition to ongoing therapy

SUMMARY:
The effect of sodium-glucose cotransporter type 2 inhibitors (SGLT2i) on the parameters of renal function in acute decompensation of chronic heart failure (ADHF) compared to standard therapy will be analyzed. Based on the dynamics of the clinical condition, the duration of hospitalization, and blood biochemical parameters (creatinine, urea, uric acid, potassium, sodium, N-terminal pro-brain natriuretic peptide - NT-proBNP) conclusions will be drawn about the possibility of using SGLT2i in this group of patients.

DETAILED DESCRIPTION:
This is a randomized multicenter prospective clinical trial involving patients over 18 years of age who were hospitalized due to decompensation of chronic heart failure (CHF).

The aim of the study is to evaluate the effect of SGLT2i on renal function in the treatment of decompensation of chronic heart failure compared to standard therapy.

The study is planned to include 370 patients with decompensated chronic heart failure. The study will be conducted in Сity clinical hospital number 7, University clinical hospital number 1.

Patients will be screened in the first 24 hours from the moment of hospitalization, inclusion and exclusion criteria will be applied. The ADHF diagnosis was made based on 1) presence of congestion (based on the presence of dyspnoea and at least two of the following:congestion on chest X-ray in straight and side projections with radiation load 0,1 mSv (СombiDiagnost R90, №2017/6644), rales on chest auscultation, peripheral edema, swelling of the cervical veins, hepatomegaly, ascites, hepatojugular reflux) 2) the need for intravenous administration of loop diuretics.

The diagnosis will be confirmed by echocardiography (ECHO) (Ge Logic F6; №9451\61287) to assess systolic (a decrease in LV ejection fraction (LVEF) <50%) and diastolic dysfunction (ratio of early diastolic transmitral E flow to the average early diastolic velocity of the fibrous ring e´ >14; left atrial volume index (LAVI) >34 ml/m2; the maximum speed of tricuspid regurgitation >2.8 m/s ( American Society of Echocardiography (ASE)/European Association of Cardiovascular Imaging (EACVI) recommendations)[11]) and the presence of an enlarged, non-collapsing on inspiration inferior vena cava (IVC).

Intravenous administration of 40 mg of furosemide (lasix; 10 mg / ml; N014865/02) is allowed no later than in the first 24 hours from the moment of admission (provided that the patient has not previously received regular loop diuretics). If prior to this hospitalization, regular therapy with loop diuretics was carried out, the daily dose should be increased by more than 2 times with the transition to intravenous administration.

During the first visit, patients who meet the inclusion criteria will be randomized by the random number table method. Participants will be divided into two groups, the main group will include patients receiving dapagliflozin (Forxiga; MP-002596) at a dose of 10 mg / day per os in addition to the current therapy. The comparison group will be patients receiving standard therapy (loop diuretics, vasodilators, digoxin, inotropic agents, vasopressors).

During the second visit (48 hours after randomization), the researcher will assess the clinical condition (blood pressure, heart rate, respiratory rate, auscultation, edema dynamics), biochemical and general blood analysis, and patient weighing in both groups of patients. Accounting for how the patient excretes fluid will be made by the research doctor by weighing in the morning on an empty stomach and calculating the volume of diuresis.

During the third visit (on the day of discharge ), the researcher will assess the clinical condition (blood pressure, heart rate, respiratory rate, auscultation, edema dynamics), biochemical and general blood analysis, and patient weighing in both groups of patients.

The criterion for acute renal injury will be an increase in serum creatinine by 0.3 mg / dl or more for 48 hours (Kidney Disease: Improving Global Outcomes (KDIGO) criteria). The criteria for refractoriness to diuretic therapy will be the need to increase the daily dose of loop diuretics by more than 2 times compared to the initial one, or the need to add another class of diuretic drugs to the therapy. (Muthiah Vaduganathan et al. Unsolved challenges in diuretic therapy for acute heart failure: a focus on diuretic response.Expert Review of Cardiovascular Therapy/ Volume 13, 2015 -Issue 10. Pages

1075-1078). The initial dose will be the daily dose of loop diuretics used on the first day of hospitalization.

In order to find out whether there were repeated hospitalizations or deaths of patients within 30 days, the study participants will be called on the 30th day after discharge.

The reliability of the differences in the groups will be determined by the Man-Whitney criterion, the differences will be considered statistically significant at p<0.05. Statistical processing of the obtained data will be carried out using the Statistical Package for the Social Sciences program version 9.0.

The study can be classified as a study of average accuracy. The significance level of 0.05 will be used as the limit of the statistical significance of the results, then according to the method of K. A. Otdelnova, the sample size of the dissertation research should be 100 observation units. The research capacity will be 80%.

ELIGIBILITY:
Inclusion criteria

1. Diagnosed ADHF (based on 1) presence of congestion (based on the presence of dyspnoea and at least two of the following:congestion on chest X-ray, rales on chest auscultation, peripheral edema, swelling of the cervical veins, hepatomegaly, ascites, hepatojugular reflux) 2) the need for intravenous administration of loop diuretics.

The diagnosis will be confirmed by echocardiography (ECHO) to assess systolic (a decrease in LV ejection fraction (LVEF) <50%) and diastolic dysfunction (ratio of early diastolic transmitral E flow to the average early diastolic velocity of the fibrous ring e´ >14; left atrial volume index (LAVI) >34 ml/m2; the maximum speed of tricuspid regurgitation >2.8 m/s ( American Society of Echocardiography (ASE)/European Association of Cardiovascular Imaging (EACVI) recommendations)[11]) and the presence of an enlarged, non-collapsing on inspiration inferior vena cava (IVC)) 2. The need for intravenous administration of loop diuretics on admission 3. Age over 18 years Patients were included after signing an informed consent Exclusion criteria

1. Cardiogenic shock (systolic blood pressure <90 mm Hg; signs of hypoperfusion (altered mental status, cold skin, diuresis <30 ml / hour, blood lactate level >2.0 mmol / l).
2. Urinary tract infection
3. Type 1 diabetes mellitus (DM1), episodes of diabetic ketoacidosis or hypoglycemia
4. Prior use of drugs from the SGLT2i group, taken regularly within 4 weeks
5. GFR<30 ml / min / 1.73 m2 (CKD-EPI).
6. Individual SGLT2i intolerance
7. Child-Pugh class C liver failure
8. Mental illness (inability to sign an informed consent, lack of understanding of possible consequences)
9. Pregnancy or breastfeeding
10. Refusal to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
death due to heart failure | through study completion, an average of 5 days
  Death during hospitalization

SECONDARY OUTCOMES:
deterioration of renal function (increase in blood creatinine by 0.3 mg / dl within 48 hours) | through study completion, an average of 5 days
  By deterioration of kidney function is meant an increase in blood creatinine by 0.3 mg / dl within 48 hours. The maximum creatinine at hospitalization, the maximum uric acid at hospitalization, an episode of hyponatremia (sodium less than 136), an episode of oligoanuria (diuresis less than 300 ml per day) will also be taken into account. Renal function will be determined at the date of inclusion and randomisation, 3-4 days of hospitalization (second visit) and the date of discharge (third visit).
development of resistance to diuretics | through study completion, an average of 5 days
  The need to increase the daily dose of loop diuretics by more than 2 times compared to the initial one, or the need to add another class of diuretic drugs to the therapy. (Muthiah Vaduganathan et al. Unsolved challenges in diuretic therapy for acute heart
  failure: a focus on diuretic response.Expert Review of Cardiovascular Therapy/ Volume 13, 2015 -Issue 10. Pages 1075-1078).
re-hospitalization about decompensation of chronic heart failure within 30 days after discharge from the hospital | up to 30 days
  30 days after discharge, patients will be called to find out whether there are repeated hospitalizations for heart failure

OTHER OUTCOMES:
weight loss during hospitalization | through study completion, an average of 5 days
  weight loss from the moment of randomization to the day of discharge
admission to the intensive care unit due to worsening heart failure during the current hospitalization | through study completion, an average of 5 days
  admission to an intensive care unit (because of hemodynamic instability, systolic blood pressure less than 90 millimeters of mercury (mm Hg.St.), severe (progressive) shortness of breath with use of additional respiratory muscles, breathing frequency more than 25\min, need for intubation, lung ventilation, the presence of symptoms of hypoperfusion, oxygen saturation less than 90% (despite oxygen therapy), brady - and tachyarrhythmias with heart rate <40 or >130 beats/min, respectively, high-
  grade atrioventricular block, life-threatening condition: acute coronary syndrome, mechanical complications of acute insufficiency of the heart valves, chest trauma, pulmonary thromboembolism, aorta dissection)

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - University Clinical Hospital number 1, Moscow
  - Сity Сlinical Нospital number 7, Moscow

IPD SHARING:
Plan to Share IPD: No
since this is prohibited by the local ethics committee

REFERENCES:
- [Background] Vaduganathan M, Kumar V, Voors AA, Butler J. Unsolved challenges in diuretic therapy for acute heart failure: a focus on diuretic response. Expert Rev Cardiovasc Ther. 2015 Oct;13(10):1075-8. doi: 10.1586/14779072.2015.1087313. Epub 2015 Sep 10. PMID 26357970
- See also: The significance level of 0.05 will be used as the limit of the statistical significance of the results, then the sample size of the research should be 100 observation units. — http://medstatistic.ru/calculators/calcsize.html